CLINICAL TRIAL: NCT03946007
Title: Quality of Life, Cognitive Function, and Physical Fitness of Melanoma and NSCLC Patients Surviving More Than 2 Years After Immune Checkpoint Inhibitor Therapy
Brief Title: Quality of Life and Physical Fitness After Immune Checkpoint Inhibitors
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201800146
Record Dates: First submitted 2018-03-05; First posted 2019-05-10 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Melanoma; Non Small Cell Lung Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — vena punction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with melanoma or NSCLC: Patients (age ≥18 years) with melanoma or NSCLC ≥2 years since treatment with at least one cycle of immune checkpoint inhibitor (CTLA-4 inhibitor, PD-(L)1 inhibitor, or both) within the Department of Medical Oncology or Pulmonary Oncology of the UMCG.

SUMMARY:
Rationale: Tremendous anti-tumor effects have been achieved using immune checkpoint inhibitors for melanoma and NSCLC with long lasting responses of more than 2 years in a substantial subgroup of patients. However, we are still largely unaware of the health-related quality of life of these patients. We should carefully and thoroughly assess the long-term burden of disease and treatment toxicity.

Objective: Primary Objective: to investigate health-related quality of life (HRQoL) of patients surviving 2 years or more after the first cycle of an immune checkpoint inhibitor for melanoma or NSCLC. Secondary Objectives: to assess neurocognitive function, endocrine function, cardiovascular risk, physical fitness, mood disorders, sexual problems, work participation in patients surviving 2 years or more after the first cycle of immune checkpoint inhibitor; to assess quality of life of the caregivers of these patients.

Study design: Observational cross-sectional study. Study population: Patients (age ≥18 years) with melanoma or NSCLC ≥2 years since treatment with at least one cycle of immune checkpoint inhibitor (CTLA-4 inhibitor, PD-(L)1 inhibitor, or both).

Main study parameters/endpoints: health-related quality of life (HRQoL) as measured using the EORTC Quality of life questionnaire (QLQ-C30). Secondary study parameters: possible late effects (neurocognitive dysfunction, endocrine disorders, dermatologic complaints, sexual disorders and infertility, increased cardiovascular risk, and fatigue), physical fitness, psychosocial issues related to work/education, mood disorders (anxiety and depression), patient and treatment-related factors potentially influencing development of late effects, well-being, and quality of life of caregivers.

DETAILED DESCRIPTION:
Participation in the study will include one study visit of approximately 2.5 hours. If possible, the study visit will be combined with a regular follow-up visit. Vena puncture is the only invasive procedure, with low risk of adverse effects. Blood will be drawn after an overnight fast. To minimize the duration of the visit, patients will be offered to fill out the questionnaires at home. Individual adverse test results will be reported to a participants' treating physician to enable treatment or follow-up as indicated. The results of the full study group will be used to guide future interventions and support for melanoma and NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with melanoma or NSCLC ≥2 years since treatment with at least one cycle of immune checkpoint inhibitor (CTLA-4 inhibitor, PD-(L)1 inhibitor, or both) within the Department of Medical Oncology or Pulmonary Oncology of the UMCG.
2. Age ≥18 years at time of immune checkpoint inhibitor treatment
3. All previous or subsequent therapies allowed, including (brain) irradiation, surgery for metastases, chemotherapy, and targeted therapy, provided stable clinical situation at time of inclusion

Exclusion Criteria:

1. Switch of systemic therapy or local antitumor intervention (surgery, radiotherapy) during last 2 months
2. Inability to understand or abide to the study protocol
3. Debilitating psychiatric illness
4. Previous treatment for malignancy other than melanoma (excluding non-melanoma skin cancer, cervical intra-epithelial neoplasia (CIN) or carcinoma in situ of breast)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An estimated 80 adult patients with advanced melanoma and 250 patients with NSCLC are treated with immune checkpoint inhibitors in the UMCG each year. Around 20% of these patients are expected to survive ≥2 years since their first cycle of immune checkpoint inhibitor. Patients will be recruited and study measurements will be performed within 3 year after start of study. We expect to include 25 melanoma and 50 NSCLC patients per treatment year.
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) | 3 years
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Core questionnaire (QLQ-C30)

SECONDARY OUTCOMES:
cognitive function | 3 years
  Hopkins Verbal Learning Test-Revised (HVLT-R);
cognitive function | 3 years
  Controlled Oral Word Association Test (COWA);
cognitive function | 3 years
  Trail Making Test (TMT)
Physical fitness | 3 years
  six-minute walk test (6MWT)
endocrine function | 3 years
  measurement of gonadal and pituitary function in blood
Quality of life of caregivers | 3 years
  Caregiver Quality of Life Index-Cancer (CQOLC)
muscle strength | 3 years
  Maximal voluntary isometric muscle force of the right and left extremity of extension of the knee, flexion of the knee, flexion of the elbow, extension of the elbow and grip-strength of the hand will be measured using a hand-held dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: J. Nuver, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands